CLINICAL TRIAL: NCT03166735
Title: A Multi-centre, Double-blind, Parallel-group, Randomised, Placebo Controlled Phase II a Study to Investigate Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of Different Doses of Orally Administered BI 1467335 During a 12-week Treatment Period Compared to Placebo in Patients With Clinical Evidence of NASH.
Brief Title: Different Doses of BI 1467335 Compared to Placebo in Patients With Clinical Evidence of NASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1386-0004; 2016-000499-83 (EudraCT Number)
Record Dates: First submitted 2017-05-24; First posted 2017-05-25 (Actual); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- BI 1467335 dose 1 (Experimental)
  Interventions: Drug: BI 1467335
- BI 1467335 dose 2 (Experimental)
  Interventions: Drug: BI 1467335
- BI 1467335 dose 3 (Experimental)
  Interventions: Drug: BI 1467335
- BI 1467335 dose 4 (Experimental)
  Interventions: Drug: BI 1467335
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1467335 — once daily
  Arms: BI 1467335 dose 1; BI 1467335 dose 2; BI 1467335 dose 3; BI 1467335 dose 4
Drug: Placebo — once daily
  Arms: Placebo

SUMMARY:
The primary objective of this study is the proof of mechanism and support of dose finding, together with the safety evaluation in patients with clinical evidence of NASH.

To gain further insight into clinical effects of AOC3 inhibition on NASH further exploratory analyses of biomarkers related to NASH and liver fibrosis will be performed. This will include the effect of BI 1467335 on reduction of secondary biomarker endpoints (ALT, AST, AP, γ-GT and CK18 fragments). Safety will be assessed throughout the study to provide key information regarding the use of BI 1467335 in patients with NASH.

ELIGIBILITY:
Inclusion criteria:

* Clinical evidence of NASH defined as a. histological evidence of NASH (no more than 3 years prior to screening) OR b. clinical imaging results suggestive of NASH (no more than 3 years prior to screening) OR within the screening phase, imaging procedures performed as per local standard) i. evidence of hepatic steatosis >5% measured by the MRI-PDFF) or assessed as moderate to severe steatosis (raised echogenicity of the liver parenchyma) by ultrasound AND ii. evidence of liver fibrosis defined as mean stiffness > 3.64 kPa as measured by the MRE protocol or mean stiffness > 7.2 kPa as measured by ultrasound based transient elastography (Fibroscan®)
* Increased ALT defined as a. ALT >1.5 ULN at screening and ALT >1.25 ULN in a local lab within 1 week to 3 months prior screening OR b. Historic ALT > 1.25 ULN more than 3 months prior to screening and two consecutive ALT > 1.5xULN must be confirmed at least 1 week apart within the screening period
* Age ≥ 18 and ≤75 years at screening
* BMI ≥25kg/m2 and <45kg/m2 at screening
* Stable body weight defined as less than 5% change in body weight in the 3 months prior to screening while being treated with the standard of care and not treated with anti-obesity medication at screening.
* Treatment with Antidiabetic concomitant medication including any insulin regimen needs to be stable for 3 months, and treatment with vitamin E needs to be stable for 6 months prior to informed consent and expected to be stable throughout the trial. All other concomitant medication has to be stable for at least 4 weeks prior screening. Concomitant medications taken to treat acute conditions (e.g. headache, sinusitis) for a short period (< 7 days) are permissible, if not otherwise prohibited.
* For female patients: Women of childbearing potential* can be randomized after a negative pregnancy test and under adequate contraception with two methods, of which at least one is highly effective, during the trial.* A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Tubal ligation is NOT a method of permanent sterilisation. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
* Signed and dated written informed consent in accordance with GCP and local legislation prior to admission to the trial.

Exclusion criteria:

* Current or history of significant alcohol consumption (defined as intake of >210g/week in males and >140g/week in females on average over a consecutive period of more than 3 months) or inability to reliably quantify alcohol consumption based on investigator judgement.
* Prior participation in an interventional NASH trial 6 months before baseline or 5 times halflife of the investigational drug, whichever is longer.
* Prior or planned bariatric surgery during study conduct, except gastric-band surgery more than 2 years prior to screening (including adjustments) with a stable body weight within the last 12 months.
* Use of drugs historically associated with liver injury, hepatic steatosis or steatohepatitis in the 4 weeks prior to screening.
* History of liver cirrhosis (fibrosis stage 4), or hepatic decompensation (e.g. ascites, hepatic encephalopathy, variceal bleeding, etc.) or history of other forms of chronic liver disease (for example Hepatitis B, Hepatitis C, autoimmune liver disease, primary biliary sclerosis, primary sclerosing cholangitis, Wilsons disease, hemochromatosis, A1At deficiency, history of liver transplantation).
* Active known chronic or relevant acute infections, such as HIV (Human Immunodeficiency Virus), \viral hepatitis, or tuberculosis. QuantiFERON® TB test and HBs Ag test will be performed during screening. Patients with a positive test result may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the patient has no evidence of active infection.
* Solid liver lesions other than haemangiomas.

  -- Suspicion or diagnosis or history of hepatocellular carcinoma (HCC)
* eGFR <60ml/min/1.73m2 at screening (CKD-EPI formula).
* ALT >5.0 ULN at screening.
* Platelet count < 150.000/μL
* Bilirubin level > ULN (except for known Gilbert´s disease with a conjugated bilirubin of < 0.3 mg/dL))
* Uncontrolled diabetes defined as an HbA1c ≥9.5% in the 3 months prior to or at screening.
* Diagnosis of a serious or unstable disease including hepatic (other than NASH), renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic , psychiatric, immunologic, or hematologic disease and other conditions that, in the clinical judgment of the investigator, are likely to interfere with the analyses of safety and efficacy in this study. Patients with an expected life expectancy of less than 2 years are also excluded.
* Major surgery (major according to the investigator's assessment) performed within 12 weeks prior to randomisation or planned during study conduct, e.g. hip replacement.
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix.
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial.
* Previous randomisation in this trial.
* Currently enrolled in another investigational device or drug study, or less than 30 days since ending another investigational device or drug study(s), or receiving other investigational treatment(s).
* Chronic drug abuse or any condition that, in the investigator's opinion, makes them an unreliable study subject or unlikely to complete the trial.
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
* Patients with Wolff-Parkinson-White Syndrome, baseline QTc > 450 ms, family history of long QT, or on medication prolonging QT time at screening or planned initiation during the trial.
* Any other clinical condition that, in the opinion of the investigator, would jeopardize patient safety while participating in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (16):
  - Southern California Research Center, Coronado, California
  - University of California San Diego, La Jolla, California
  - eStudySite, La Mesa, California
  - National Research Institute, Los Angeles, California
  - Quest Clinical Research, San Francisco, California
  - Florida Research Institute, Lakewood Rch, Florida
  - Genoma Research Group, Inc, Miami, Florida
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Northwell Health, Manhasset, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Diabetes and Endocrinology Consultants, PC, Morehead City, North Carolina
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - Pinnacle Clinical Research, Live Oak, Texas
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Belgium (4):
  - Edegem - UNIV UZ Antwerpen, Edegem
  - AZ Maria Middelares, Ghent
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Toronto Liver Centre, Toronto, Ontario
- France (2):
  - HOP Claude Huriez, Lille
  - HOP La Pitié Salpêtrière, Paris
- Germany (6):
  - Universitätsklinikum Aachen, AöR, Aachen
  - Universitätsklinikum Köln (AöR), Cologne
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Würzburg, Würzburg
- St James's Hospital, Dublin, Ireland
- Netherlands (3):
  - Amsterdam UMC, Locatie AMC, Amsterdam
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Radboud Universitair Medisch Centrum, Nijmegen
- Spain (5):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Virgen del Rocío, Seville
  - Hospital General Universitario de Valencia, Valencia
- United Kingdom (4):
  - Queen Elizabeth Hospital, Birmingham
  - Aintree University Hospital, Liverpool
  - Manchester Royal Infirmary, Manchester
  - Royal Stoke University Hospital, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Newsome PN, Sanyal AJ, Neff G, Schattenberg JM, Ratziu V, Ertle J, Link J, Mackie A, Schoelch C, Lawitz E; BI 1467335 NASH Phase IIa trial team. A randomised Phase IIa trial of amine oxidase copper-containing 3 (AOC3) inhibitor BI 1467335 in adults with non-alcoholic steatohepatitis. Nat Commun. 2023 Nov 6;14(1):7151. doi: 10.1038/s41467-023-42398-w. PMID 37932258
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is a multi-centre, double-blind, parallel-group, randomised, placebo-controlled phase IIa study to investigate safety, tolerability, pharmacodynamics, and pharmacokinetics of different doses of orally administered BI 1467335 (for 12-weeks) compared to placebo in patients with clinical evidence of Non-alcoholic steato-hepatitis (NASH).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Placebo: Matching placebo taken daily for 12 weeks. Tablets taken orally with water in the morning, fasted, 1 hour before breakfast. Film-coated placebo tablets were supplied. For blinding reasons, all patients took 5 tablets placebo daily.
- BI 1467335 1 Milligram (mg): 1 milligram (mg) BI 1467335 taken daily for 12 weeks. Tablets taken orally with water in the morning, fasted, 1 hour before breakfast. Film-coated tablets were supplied as 1 mg and 5 mg dose strengths. For blinding reasons, all patients took 5 tablets verum or placebo daily.
- BI 1467335 3 Milligram (mg): 3 milligram (mg) BI 1467335 taken daily for 12 weeks. Tablets taken orally with water in the morning, fasted, 1 hour before breakfast. Film-coated tablets were supplied as 1 mg and 5 mg dose strengths. For blinding reasons, all patients took 5 tablets verum or placebo daily.
- BI 1467335 6 Milligram (mg): 6 milligram (mg) BI 1467335 taken daily for 12 weeks. Tablets taken orally with water in the morning, fasted, 1 hour before breakfast. Film-coated tablets were supplied as 1 mg and 5 mg dose strengths. For blinding reasons, all patients took 5 tablets verum or placebo daily.
- BI 1467335 10 Milligram (mg): 10 milligram (mg) BI 1467335 taken daily for 12 weeks. Tablets taken orally with water in the morning, fasted, 1 hour before breakfast. Film-coated tablets were supplied as 1 mg and 5 mg dose strengths. For blinding reasons, all patients took 5 tablets verum or placebo daily.
Period: Overall Study
Arm/Group | Placebo | BI 1467335 1 Milligram (mg) | BI 1467335 3 Milligram (mg) | BI 1467335 6 Milligram (mg) | BI 1467335 10 Milligram (mg)
Started | 33 | 16 | 16 | 17 | 32
Treated | 32 | 16 | 16 | 17 | 32
Completed | 32 | 13 | 13 | 16 | 28
Not Completed | 1 | 3 | 3 | 1 | 4
Not completed — Not Treated | 1 | 0 | 0 | 0 | 0
Not completed — follow-up not completed as planned | 0 | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 2
Not completed — Lost to Follow-up | 0 | 2 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): all patients who signed the informed consent and were treated with at least one dose of the trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI 1467335 1 Milligram (mg) | BI 1467335 3 Milligram (mg) | BI 1467335 6 Milligram (mg) | BI 1467335 10 Milligram (mg) | Total
Number analyzed (Participants) | 32 | 16 | 16 | 17 | 32 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (12.3) | 52.6 (13.3) | 53.9 (11.5) | 48.2 (10.1) | 49.8 (14.0) | 51.1 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 8 | 9 | 18 | 58
  Male | 19 | 6 | 8 | 8 | 14 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 5 | 5 | 4 | 8 | 33
  Not Hispanic or Latino | 21 | 11 | 11 | 13 | 24 | 80
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 0 | 0 | 2
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 30 | 14 | 16 | 17 | 32 | 109
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Plasma amine oxidase copper-containing 3 (AOC3) baseline concentration [Mean (Standard Deviation); unit: microgram per liter (µg/l)] — Plasma amine oxidase copper-containing 3 (AOC3) baseline concentration Population: Treated Set (TS): all patients who signed the informed consent and were treated with at least one dose of the trial medication.
  For 3 patients no AOC3 baseline data was collected.
  microgram per liter (µg/l)
    number analyzed (Participants) | 32 | 14 | 16 | 17 | 31 | 110
    (all) | 471.4063 (165.6802) | 537.7143 (204.4100) | 498.0000 (141.0225) | 527.2941 (142.3722) | 516.1613 (144.0727) | 504.9636 (157.4936)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Amine Oxidase Copper-containing 3 (AOC3) Activity After 12 Weeks of Treatment, Relative to Baseline in Percent
Description: The patient-specific plasma AOC3 activity at time t (24 hours after the last dose in week 12) relative to baseline in percentage was calculated as follows:
  %AOC3at = [(AOC3at - AOC3at,back) ⁄ (AOC3abase - AOC3abase,back)]*100
  With AOC3at the AOC3 activity measured at time t, AOC3at,back the background noise at time t, AOC3abase the AOC3 activity measured at baseline and AOC3abase,back the background noise at baseline.
  A dose-response relationship was analysed using a non-linear regression model to estimate the daily dosage needed to reach 10% of AOC3 activity (i.e. 90% inhibition) 12 weeks after treatment.
Time Frame: Day 1 (baseline), day 15, 29, 43, 57 and 85 (time t) 24 hours after the last dose of BI 1467335.
Population: Per Protocol Set (PPS): Patients who signed informed consent, were treated with at least one dose of the trial medication, without any important protocol deviations leading to exclusion and who had non-missing baseline and at least one non-missing post-baseline and on-treatment measurement on any primary, secondary or further biomarker endpoint.
Measure: Mean (Standard Deviation); unit: Percentage relative to baseline
Arm/Group | Placebo | BI 1467335 1 Milligram (mg) | BI 1467335 3 Milligram (mg) | BI 1467335 6 Milligram (mg) | BI 1467335 10 Milligram (mg)
Number analyzed (Participants) | 30 | 12 | 14 | 11 | 24
Percentage relative to baseline | 102 (13.0) | 24.0 (11.9) | 13.1 (10.4) | 8.27 (5.19) | 2.06 (3.62)
Statistical Analysis 1: Comparison: Placebo vs BI 1467335 1 Milligram (mg) vs BI 1467335 3 Milligram (mg) vs BI 1467335 6 Milligram (mg) vs BI 1467335 10 Milligram (mg); D10: Estimated dose reaching <=10% activity the first time; Test type: Other; non-linear regression; Predicted mean daily dose in mg = 3.45, Standard Error of Mean 0.10 — The model fit used power of mean variance estimates (POM) to account for heterogeneity

2. Secondary Outcome: Percentage of Participants With Drug-related Adverse Events (AEs)
Description: Percentage of participants with drug-related adverse events (AEs). Percentages are calculated using total number of patients per treatment as the denominator.
Time Frame: Start of treatment till end of treatment + 28 days, up to 113 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | BI 1467335 1 Milligram (mg) | BI 1467335 3 Milligram (mg) | BI 1467335 6 Milligram (mg) | BI 1467335 10 Milligram (mg)
Number analyzed (Participants) | 32 | 16 | 16 | 17 | 32
Percentage of participants | 25.0 | 31.3 | 12.5 | 11.8 | 25.0

3. Secondary Outcome: Alanine Aminotransaminase (ALT) After 12 Weeks of Treatment, Relative to Baseline in Percent
Description: Alanine aminotransaminase (ALT) after 12 weeks of treatment, relative to baseline in percent. Number analyzed lower than N in PPS if there is missing data for specific timepoints.
  The unit of measure is: percentage relative to baseline = [post baseline (time t)/baseline]*100%
  Statistical analyses description: A Mixed effects Model for Repeated Measurements (MMRM) over time including fixed effects for 'base', 'treatment', 'time', 'base*time' interaction, and 'treatment*time' interaction was performed. The MMRM estimates for the treatment effects at Week 12 and the corresponding covariance matrix were used to analyse the dose-response relationship using the Multiple contrast test (MCPMod). A test for non-flat dose-response relationship was first performed. If this relationship could be shown, the best fitting model out of a set of candidate models (Sigmoidal Emax, Logistic, Quadratic, Linear, Exponential, Linear logistic, Emax and Betamod) was to be selected and fitted.
Time Frame: Day 1 (baseline), day 15, 29, 43, 57 and 85 (time t) 24 hours after the last dose of BI 1467335.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percentage relative to baseline
Arm/Group | Placebo | BI 1467335 1 Milligram (mg) | BI 1467335 3 Milligram (mg) | BI 1467335 6 Milligram (mg) | BI 1467335 10 Milligram (mg)
Number analyzed (Participants) | 28 | 12 | 13 | 14 | 27
Percentage relative to baseline | 92.66 (106.55) | 97.32 (110.13) | 87.49 (109.79) | 80.61 (109.43) | 77.57 (106.66)
Statistical Analysis 1: Comparison: Placebo vs BI 1467335 1 Milligram (mg) vs BI 1467335 3 Milligram (mg) vs BI 1467335 6 Milligram (mg) vs BI 1467335 10 Milligram (mg); Test type: Other — The MMRM included fixed effects for 'base', 'treatment', 'time', 'base*time' interaction, and 'treatment*time' interaction. Estimates were used to test dose-response relationship using MCPMod; p = 0.0212, MCPMod Sigmoidal Emax model fit. — p<0.05 is a significant test result (rejecting the null hypothesis of a flat dose-response curve) with alpha 0.05, one-sided; 30% of the maximum effect is achieved at 3 mg and 90% of the maximum effect is achieved at 7 mg of BI 1467335

4. Secondary Outcome: Aspartate Aminotransferase (AST) After 12 Weeks of Treatment, Relative to Baseline in Percent
Description: Aspartate aminotransferase (AST) after 12 weeks of treatment, relative to baseline in percent. Number analyzed lower than N in PPS if there is missing data for specific timepoints.
  The unit of measure is: percentage relative to baseline = [post baseline (time t)/baseline]*100%
  Statistical analyses description: A Mixed effects Model for Repeated Measurements (MMRM) over time including fixed effects for 'base', 'treatment', 'time', 'base*time' interaction, and 'treatment*time' interaction was performed. The MMRM estimates for the treatment effects at Week 12 and the corresponding covariance matrix were used to analyse the dose-response relationship using the Multiple contrast test (MCPMod). A test for non-flat dose-response relationship was first performed. If this relationship could be shown, the best fitting model out of a set of candidate models (Sigmoidal Emax, Logistic, Quadratic, Linear, Exponential, Linear logistic, Emax and Betamod) was to be selected and fitted.
Time Frame: Day 1 (baseline), day 15, 29, 43, 57 and 85 (time t) 24 hours after the last dose of BI 1467335.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percentage relative to baseline
Arm/Group | Placebo | BI 1467335 1 Milligram (mg) | BI 1467335 3 Milligram (mg) | BI 1467335 6 Milligram (mg) | BI 1467335 10 Milligram (mg)
Number analyzed (Participants) | 27 | 12 | 13 | 14 | 23
Percentage relative to baseline | 93.77 (105.91) | 105.17 (108.93) | 90.09 (108.72) | 84.12 (108.34) | 87.83 (106.26)
Statistical Analysis 1: Comparison: Placebo vs BI 1467335 1 Milligram (mg) vs BI 1467335 3 Milligram (mg) vs BI 1467335 6 Milligram (mg) vs BI 1467335 10 Milligram (mg); Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.1270, MCPMod Sigmoidal Emax model fit. — [p-value comment as in outcome 3, analysis 1]; 30% of the maximum effect is achieved at 3 mg and 90% of the maximum effect is achieved at 7 mg of BI 1467335

5. Secondary Outcome: Alkaline Phosphatase (AP) After 12 Weeks of Treatment, Relative to Baseline in Percent
Description: Alkaline phosphatase (AP) after 12 weeks of treatment, relative to baseline in percent. Number analyzed lower than N in PPS if there is missing data for specific timepoints.
  The unit of measure is: percentage relative to baseline = [post baseline (time t)/baseline]*100%
  Statistical analyses description: A Mixed effects Model for Repeated Measurements (MMRM) over time including fixed effects for 'base', 'treatment', 'time', 'base*time' interaction, and 'treatment*time' interaction was performed. The MMRM estimates for the treatment effects at Week 12 and the corresponding covariance matrix were used to analyse the dose-response relationship using the Multiple contrast test (MCPMod). A test for non-flat dose-response relationship was first performed. If this relationship could be shown, the best fitting model out of a set of candidate models (Sigmoidal Emax, Logistic, Quadratic, Linear, Exponential, Linear logistic, Emax and Betamod) was to be selected and fitted.
Time Frame: Day 1 (baseline), day 15, 29, 43, 57 and 85 (time t) 24 hours after the last dose of BI 1467335.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percentage relative to baseline
Arm/Group | Placebo | BI 1467335 1 Milligram (mg) | BI 1467335 3 Milligram (mg) | BI 1467335 6 Milligram (mg) | BI 1467335 10 Milligram (mg)
Number analyzed (Participants) | 29 | 12 | 13 | 14 | 28
Percentage relative to baseline | 96.62 (102.31) | 97.58 (103.56) | 100.52 (103.45) | 98.47 (103.34) | 94.71 (102.34)
Statistical Analysis 1: Comparison: Placebo vs BI 1467335 1 Milligram (mg) vs BI 1467335 3 Milligram (mg) vs BI 1467335 6 Milligram (mg) vs BI 1467335 10 Milligram (mg); Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.3324, MCPMod exponential model fit. — [p-value comment as in outcome 3, analysis 1]; 90% of the maximum effect is achieved at 7 mg of BI 1467335

6. Secondary Outcome: Gamma-glutamyltransferase (GGT) After 12 Weeks of Treatment, Relative to Baseline in Percent
Description: Gamma-glutamyltransferase (GGT) after 12 weeks of treatment, relative to baseline in percent. Number analyzed lower than N in PPS if there is missing data for specific timepoints.
  The unit of measure is: percentage relative to baseline = [post baseline (time t)/baseline]*100%
  Statistical analyses description: A Mixed effects Model for Repeated Measurements (MMRM) over time including fixed effects for 'base', 'treatment', 'time', 'base*time' interaction, and 'treatment*time' interaction was performed. The MMRM estimates for the treatment effects at Week 12 and the corresponding covariance matrix were used to analyse the dose-response relationship using the Multiple contrast test (MCPMod). A test for non-flat dose-response relationship was first performed. If this relationship could be shown, the best fitting model out of a set of candidate models (Sigmoidal Emax, Logistic, Quadratic, Linear, Exponential, Linear logistic, Emax and Betamod) was to be selected and fitted.
Time Frame: Day 1 (baseline), day 15, 29, 43, 57 and 85 (time t) 24 hours after the last dose of BI 1467335.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percentage relative to baseline
Arm/Group | Placebo | BI 1467335 1 Milligram (mg) | BI 1467335 3 Milligram (mg) | BI 1467335 6 Milligram (mg) | BI 1467335 10 Milligram (mg)
Number analyzed (Participants) | 29 | 12 | 13 | 14 | 28
Percentage relative to baseline | 91.37 (105.24) | 99.42 (108.25) | 92.44 (108.09) | 99.51 (107.71) | 83.70 (105.40)
Statistical Analysis 1: Comparison: Placebo vs BI 1467335 1 Milligram (mg) vs BI 1467335 3 Milligram (mg) vs BI 1467335 6 Milligram (mg) vs BI 1467335 10 Milligram (mg); Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.1290, MCPMod exponential model fit. — [p-value comment as in outcome 3, analysis 1]; 90% of the maximum effect is achieved at 7 mg of BI 1467335

7. Secondary Outcome: Caspase-cleaved Cytokeratin 18 (CK-18 Caspase) After 12 Weeks of Treatment, Relative to Baseline in Percent
Description: Caspase-cleaved cytokeratin 18 (CK-18 caspase) after 12 weeks of treatment, relative to baseline in percent. Number analyzed lower than N in PPS if there is missing data for specific timepoints.
  The unit of measure is: percentage relative to baseline = [post baseline (time t)/baseline]*100%
  Statistical analyses description: A MMRM over time including fixed effects for 'base', 'treatment', 'time', 'base*time' interaction, and 'treatment*time' interaction was performed. The MMRM estimates for the treatment effects at Week 12 and the corresponding covariance matrix were used to analyse the dose-response relationship using the Multiple contrast test (MCPMod). A test for non-flat dose-response relationship was first performed. If this relationship could be shown, the best fitting model out of a set of candidate models (Sigmoidal Emax, Logistic, Quadratic, Linear, Exponential, Linear logistic, Emax and Betamod) was to be selected and fitted.
Time Frame: Day 1 (baseline), day 15, 29, 43, 57 and 85 (time t) 24 hours after the last dose of BI 1467335.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percentage relative to baseline
Arm/Group | Placebo | BI 1467335 1 Milligram (mg) | BI 1467335 3 Milligram (mg) | BI 1467335 6 Milligram (mg) | BI 1467335 10 Milligram (mg)
Number analyzed (Participants) | 29 | 12 | 12 | 14 | 26
Percentage relative to baseline | 101.35 (111.15) | 155.04 (117.61) | 96.87 (117.54) | 80.51 (116.32) | 78.08 (111.59)
Statistical Analysis 1: Comparison: Placebo vs BI 1467335 1 Milligram (mg) vs BI 1467335 3 Milligram (mg) vs BI 1467335 6 Milligram (mg) vs BI 1467335 10 Milligram (mg); Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.0042, MCPMod Sigmoidal Emax model fit. — [p-value comment as in outcome 3, analysis 1]; 30% of the maximum effect is achieved at 3 mg and 90% of the maximum effect is achieved at 7 mg of BI 1467335

8. Secondary Outcome: Total Cytokeratin 18 (CK-18 Total) After 12 Weeks of Treatment, Relative to Baseline in Percent
Description: Total cytokeratin 18 (CK-18 total) after 12 weeks of treatment, relative to baseline in percent. Number analyzed lower than N in PPS if there is missing data for specific timepoints.
  The unit of measure is: percentage relative to baseline = [post baseline (time t)/baseline]*100%.
  Statistical analyses description: A Mixed effects Model for Repeated Measurements (MMRM) over time including fixed effects for 'base', 'treatment', 'time', 'base*time' interaction, and 'treatment*time' interaction was performed. The MMRM estimates for the treatment effects at Week 12 and the corresponding covariance matrix were used to analyse the dose-response relationship using the Multiple contrast test (MCPMod). A test for non-flat dose-response relationship was first performed. If this relationship could be shown, the best fitting model out of a set of candidate models (Sigmoidal Emax, Logistic, Quadratic, Linear, Exponential, Linear logistic, Emax and Betamod) was to be selected and fitted.
Time Frame: Day 1 (baseline), day 15, 29, 43, 57 and 85 (time t) 24 hours after the last dose of BI 1467335.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percentage relative to baseline
Arm/Group | Placebo | BI 1467335 1 Milligram (mg) | BI 1467335 3 Milligram (mg) | BI 1467335 6 Milligram (mg) | BI 1467335 10 Milligram (mg)
Number analyzed (Participants) | 28 | 11 | 13 | 14 | 26
Percentage relative to baseline | 92.44 (109.13) | 128.33 (114.64) | 99.56 (113.78) | 94.74 (113.10) | 81.47 (109.35)
Statistical Analysis 1: Comparison: Placebo vs BI 1467335 1 Milligram (mg) vs BI 1467335 3 Milligram (mg) vs BI 1467335 6 Milligram (mg) vs BI 1467335 10 Milligram (mg); Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.0728, MCPMod exponential model fit. — [p-value comment as in outcome 3, analysis 1]; 90% of the maximum effect is achieved at 7 mg of BI 1467335

ADVERSE EVENTS:
Time Frame: start of treatment till end of treatment + 28 days, up to 113 days.
Description: Adverse events are reported based on the Treated Set (all patients who signed the informed consent and were treated with at least one dose of the trial medication).
Groups:
- Total BI 1467335: All participant who took a dose of BI 1467335.
Arm/Group | Placebo | BI 1467335 1 Milligram (mg) | BI 1467335 3 Milligram (mg) | BI 1467335 6 Milligram (mg) | BI 1467335 10 Milligram (mg) | Total BI 1467335
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/16 | 0/16 | 0/17 | 0/32 | 0/81
Serious Adverse Events (participants affected / at risk) | 1/32 | 1/16 | 1/16 | 0/17 | 0/32 | 2/81
Other Adverse Events (participants affected / at risk) | 18/32 | 12/16 | 12/16 | 13/17 | 17/32 | 54/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=32) | BI 1467335 1 Milligram (mg) (N=16) | BI 1467335 3 Milligram (mg) (N=16) | BI 1467335 6 Milligram (mg) (N=17) | BI 1467335 10 Milligram (mg) (N=32) | Total BI 1467335 (N=81)
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=32) | BI 1467335 1 Milligram (mg) (N=16) | BI 1467335 3 Milligram (mg) (N=16) | BI 1467335 6 Milligram (mg) (N=17) | BI 1467335 10 Milligram (mg) (N=32) | Total BI 1467335 (N=81)
Vertigo (Ear and labyrinth disorders) | 2 | 1 | 0 | 0 | 1 | 2
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1 | 2 | 3 | 7
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2 | 3
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 4 | 1 | 0 | 5 | 10
Pouchitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Early satiety (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 3 | 0 | 1 | 0 | 5 | 6
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 2
Hepatic pain (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 1 | 1 | 3
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 1
Gastroenteritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 3 | 3 | 2 | 1 | 5 | 11
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 2
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 2 | 0 | 0 | 1 | 3
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 2
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 2
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 1 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 2
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 0 | 3 | 6
Headache (Nervous system disorders) | 4 | 3 | 0 | 4 | 2 | 9
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 2
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 1
Subclavian steal syndrome (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Global Amendment 5 (dated 12 Sep 2018): Sample size reduction from 147 to 108 randomised patients due to a lower expected variability for ALT based on new external and blinded internal data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT03166735/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT03166735/SAP_001.pdf